CLINICAL TRIAL: NCT02203279
Title: Evaluation of Three Hard Relining Materials in Complete Dentures: An In-vivo Study
Brief Title: Evaluation of Three Hard Relining Materials in Complete Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-RemPro-02-2014
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Complete Mandibular Dentures With Poor Retention
Keywords: Chair-side hard relining; complete denture; patients' satisfaction; supporting tissues; autopolymerized reline resins; heat cured relining material
MeSH Terms: interventions — tokuyama rebase fast II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rebase II Fast (Experimental): The direct chair-side relining materiel 'Rebase II Fast' will be used.
  Interventions: Other: Rebase II Fast
- Flexacryl (Experimental): The direct chair-side relining material Flexacryl will be used
  Interventions: Other: Flexacryl
- Vertex (Experimental): Vertex is a heat-cured resin material which is going to be used for indirect relining
  Interventions: Other: Vertex

INTERVENTIONS:
Other: Rebase II Fast — It is going to be used a direct relining material
  Arms: Rebase II Fast
Other: Flexacryl — This is going to be used as a second direct relining material
  Arms: Flexacryl
Other: Vertex — This is going to be used as an indirect relining material
  Arms: Vertex

SUMMARY:
Purpose: The purpose of this study is to evaluate three hard relining materials after 3 and 6 months of use with mandibular complete dentures. The effect of hard relining materials on supporting tissues and patients' satisfaction will also be assessed.

Materials and Methods: 36 complete edentulous patients who already have maxillary dentures and complaining of instable mandibular dentures will be invited to participate in this study. Mandibular dentures will be relined randomly by one of three relining materials: two chairside relining materials (Tokuyama Rebase II Fast, Tokuyama Dental Co, Japan), and (Flexacryl Hard, Lang Co, USA) and one heat cured acrylic resin (Vertex, Dental technology Co, Holland).

The color stability of relining material, peeling, and the effect on supporting tissue will be assessed by two separate prosthodontists after 3 and 6 months of follow up. In addition, patients will be asked to grade there overall satisfaction on a Visual Analogue Scale (VAS) ranging from 0 to 100.

DETAILED DESCRIPTION:
Relining denture is a process of resurfacing the tissue side of a denture to make it fit more accurately Direct relining of removable dentures with hard chair-side reline materials is suitable for improving the fit of the denture bases to the supporting tissues. Chairside reline materials are more convenient than those processed in a laboratory because the direct method is faster and does not cause clinically significant dimensional changes of the reline resin. However, when autopolymerized reline resins are used with a direct method, several problems can occur as burning sensation caused by monomers, an exothermic heat reaction and an unpleasant odor.

There are three types of hard relining chair-side materials: Dual-polymerized Visible light-polymerized as Triad DuaLine, Light Liner (Hard), Astron LC (Hard).Visible light-polymerized as Lightdon-U, Triad Hi-Flow Reline Material, Triad VLC Reline Material. Finally, autopolymerized as New Truline, Tokuyama Rebase II (Fast) , GC Reline. Other concerns related to direct reline materials include patient tolerance (taste, temperature, odor), color stability, durability and ease of handling and polishing.

Few studies evaluated the effect of disinfection solutions on relining materials properties as roughness and hardness. In one study, disinfectant solutions caused a decrease in hardness, whereas with roughness, the materials tested showed a statistically significant increase, except for Tokuyama. Depending on the examined relining materials, some materials have increased and the others have decreased surface roughness after immersion in disinfecting solutions or microwave disinfection.

All previous laboratory studies concentrated on the effects of disinfection on relining materials properties as roughness, hardness, color change. However, the clinical studies did not compare chemically cured and heat cured relining materials and their effects on supporting tissue. The aim of this study is to evaluate the clinical performance of two -chemically cured- and heat cured denture relining material after 3 and 6 months of use. In addition, the effect of hard relining materials on supporting tissues, and patients' satisfaction has not been evaluated yet.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45-80 year,
* complete maxillary and lower dentures
* Mandibular dentures with poor retention

Exclusion Criteria:

* Patients with good stability of mandibular dentures.
* Partial maxillary edentulous patients

Ages: 47 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Supporting Alveolar Mucosa Status_3 | This will be measured at three months following relining
  According to a clinical examination by two prosthodontists, the supporting alveolar mucosa will be given one of the following levels:
  Class I: The presence of reddish soft tissues extending to more than half of the area of the supporting mucosa or the presence of large areas of movable tissues.
  Class II: The presence of irritated soft tissues extending to about third of the area of the supporting mucose or the presence of some areas of movable tissues at the top of the alveolar ridge.
  Class III: The soft tissues appear in general as normal and fixed except for small isolated areas.
  Class IV: The soft tissues appear normal and fixed without any signs of irritation or denture-induced injuries.
Supporting Alveolar Mucosa Status_6 | This variable will be assessed at six months following relining
  According to a clinical examination by two prosthodontists, the supporting alveolar mucosa will be given one of the following levels:
  Class I: The presence of reddish soft tissues extending to more than half of the area of the supporting mucosa or the presence of large areas of movable tissues.
  Class II: The presence of irritated soft tissues extending to about third of the area of the supporting mucose or the presence of some areas of movable tissues at the top of the alveolar ridge.
  Class III: The soft tissues appear in general as normal and fixed except for small isolated areas.
  Class IV: The soft tissues appear normal and fixed without any signs of irritation or denture-induced injuries.
Color Stability_3 | This will be assessed at three moths following relining
  The color stability variable has four degrees on clinical examination:
  1. no change
  2. simple
  3. medium
  4. large

SECONDARY OUTCOMES:
Color Stability_6 | This be assessed at six months following relining
  The color stability variable has four degrees on clinical examination:
  no change simple medium large
Peeling_3 | This variable is going to be assessed at three months following relining
  This variable is going to be inspected clinically and it has two categories:
  1. peeling more than 4 mm
  2. peeling less than 4 mm
Peeling_6 | This variable is going to be assessed at six months following relining
  This variable is going to be inspected clinically and it has two categories:
  1. peeling more than 4 mm
  2. peeling less than 4 mm
Satisfaction_3 | This is going to be measured at three months following relining
  Patient's satisfaction: patients will be asked to grade there overall satisfaction on a visual analogue scale (VAS) ranging from 0 to 100.
Satisfaction_6 | This is going to be measured at six months following relining
  Patient's satisfaction: patients will be asked to grade there overall satisfaction on a visual analogue scale (VAS) ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Teriaky, DDS MSc, Principal Investigator — PhD student, Department of Removable Prosthodontics, University of Damascus Dental School, Damascus; Muhannad Alssadi, DDS MSc PhD, Study Director — Associate Professor, Removable Prosthodontics Department, University of Damascus Dental School, Damascus
Locations (1):
- Department of Removable Prosthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Al Rifaiy MQ. Shear bond strength between light polymerized hard reline resin and denture base resin subjected to long term water immersion. Saudi Dent J. 2012 Jan;24(1):23-7. doi: 10.1016/j.sdentj.2011.10.004. Epub 2011 Nov 20. PMID 23960524
- [Background] Arima T, Murata H, Hamada T. Analysis of composition and structure of hard autopolymerizing reline resins. J Oral Rehabil. 1996 May;23(5):346-52. doi: 10.1111/j.1365-2842.1996.tb00863.x. PMID 8736448
- [Background] Pinto Lde R, Acosta EJ, Tavora FF, da Silva PM, Porto VC. Effect of repeated cycles of chemical disinfection on the roughness and hardness of hard reline acrylic resins. Gerodontology. 2010 Jun;27(2):147-53. doi: 10.1111/j.1741-2358.2009.00282.x. Epub 2009 Jun 8. PMID 19508322
- [Background] Haywood J, Basker RM, Watson CJ, Wood DJ. A comparison of three hard chairside denture reline materials. Part I. Clinical evaluation. Eur J Prosthodont Restor Dent. 2003 Dec;11(4):157-63. PMID 14737792
- [Background] Hong G, Murata H, Li Y, Sadamori S, Hamada T. Influence of denture cleansers on the color stability of three types of denture base acrylic resin. J Prosthet Dent. 2009 Mar;101(3):205-13. doi: 10.1016/S0022-3913(09)60032-9. PMID 19231574
- [Background] Machado AL, Breeding LC, Vergani CE, da Cruz Perez LE. Hardness and surface roughness of reline and denture base acrylic resins after repeated disinfection procedures. J Prosthet Dent. 2009 Aug;102(2):115-22. doi: 10.1016/S0022-3913(09)60120-7. PMID 19643225
- [Background] Machado AL, Giampaolo ET, Vergani CE, Souza JF, Jorge JH. Changes in roughness of denture base and reline materials by chemical disinfection or microwave irradiation: surface roughness of denture base and reline materials. J Appl Oral Sci. 2011 Oct;19(5):521-8. doi: 10.1590/s1678-77572011000500015. PMID 21986658
- [Background] Matsumura H, Tanoue N, Kawasaki K, Atsuta M. Clinical evaluation of a chemically cured hard denture relining material. J Oral Rehabil. 2001 Jul;28(7):640-4. doi: 10.1046/j.1365-2842.2001.00701.x. PMID 11422696
- [Background] Murata H, Seo RS, Hamada T, Polyzois GL, Frangou MJ. Dynamic mechanical properties of hard, direct denture reline resins. J Prosthet Dent. 2007 Oct;98(4):319-26. doi: 10.1016/S0022-3913(07)60105-X. PMID 17936130
- [Background] Ogle RE, Sorensen SE, Lewis EA. A new visible light-cured resin system applied to removable prosthodontics. J Prosthet Dent. 1986 Oct;56(4):497-506. doi: 10.1016/0022-3913(86)90397-5. PMID 3463760
- [Background] Wyatt CC, Harrop TJ, MacEntee MI. A comparison of physical characteristics of six hard denture reline materials. J Prosthet Dent. 1986 Mar;55(3):343-6. doi: 10.1016/0022-3913(86)90117-4. PMID 3457166